CLINICAL TRIAL: NCT05522933
Title: Development and Evaluation of an Online Multidimensional Musculoskeletal Health Promotion Program for Low-skilled Workers in the Low-Income Community in Covid-19 Pandemic Situation - a Feasibility Study
Brief Title: Development and Evaluation of an Online Multidimensional Musculoskeletal Health Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSEARS20220624001
Record Dates: First submitted 2022-08-22; First posted 2022-08-31 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2022-08

CONDITIONS: Occupational Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Musculoskeletal Health (Experimental): The intervention group will receive the 4 weekly workshops
  Interventions: Other: 4 weekly musculoskeletal health promotion workshops with stretching and muscle-strengthening exercise

INTERVENTIONS:
Other: 4 weekly musculoskeletal health promotion workshops with stretching and muscle-strengthening exercise — The modified online multidimensional musculoskeletal health promotion program will consist of 4 weekly workshops for 90-minute each for a group size of 8-12 participants. The topics of the workshop are: (1) exercise and health & work; (2) prevention of musculoskeletal problems; (3) musculoskeletal health and traditional Chinese medicine; and (4) mental health and community resources. Each workshop will consist of stretching and muscle strengthening exercises (30 minutes), a health education topic (about 45 minutes), and a question-and-answer period (about 15 minutes).

SUMMARY:
Globally, work-related musculoskeletal symptoms (WRMSs) have become one of the major public health issues, with musculoskeletal problems contributing to the largest proportion of lost work productivity. Literature has reported that grassroots working-class workers (also known as low-skilled workers) are the most vulnerable group to WRMSs as their work mostly exposes them to the identified risk factors. However, not many intervention studies have been conducted for low-skilled workers to prevent WRMSs.

Based on the concept of the multidimensional approach from the literature, and the project team's previous evidence-based research results, this project will modify the project team's face-to-face evidence-based musculoskeletal health promotion program to an online mode with 4 weekly 45-minute workshops for low-skilled workers in the community under the Covid-19 pandemic situation. Thus, the project has the following specific objectives:

(i) To determine the feasibility of conducting the proposed online program (ii) To examine the acceptability and satisfaction of the online program from the workers' perspectives (iii) To evaluate the potential effects of the online program on the primary outcomes: compliance with exercise regimes, improvement of musculoskeletal literacy, and reduction of the number of body parts with WRMSs (iv) To evaluate the potential effects of the online program on the secondary outcomes: reduction of adverse workstyle, improvement of exercise self-efficacy, mental health, body mass index, hip-waist ratio, and blood pressure measurements

ELIGIBILITY:
Inclusion Criteria:

* low-skilled workers aged ≥ 18
* working full-time or part-time,
* with at least one body part that had been affected by WRMSs for at least one month.

Exclusion Criteria:

* engagement in WRMS prevention programs in the workplace at the time of the study,
* undergoing medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Compliance with exercise regimes | Change from the measurement at baseline (T0) to one week after intervention (T1)
  Exercise regimes will be measured by number of times the participant perform the exercise taught. The higher the number represents a better outcome
Musculoskeletal literacy | Change from the measurement at baseline (T0) to one week after intervention (T1)
  Musculoskeletal literacy will be measured by a scale with 25 items with right or wrong answer. Score 1 will be denoted to right answer while score 0 will be denoted to wrong answer. Thus, the higher the score represents a better outcome
Incidence of body parts with work-related musculoskeletal systems (WRMSs) | Change from the measurement at baseline (T0) to one week after intervention (T1)
  The incidence of body parts with WRMSs will be measured by a modified general Nordic Musculoskeletal questionnaire to collect data about pain, aches or discomfort in different body parts. Score 1 will be denoted to one body part with WRMSs and Score 0 will be denoted to the body part without WRMSs. Thus, the higher the score represents a worse outcome.

SECONDARY OUTCOMES:
Adverse workstyle | Change from the measurement at baseline (T0) to one week after intervention (T1)
  Adverse workstyle will be measured by a 24-item Chinese Workstyle Short Form for WRMSs with a 5-point Likert scale (0 = almost never and 4 = almost always). It consists of 4 subscales: work through pain (6 items), social reactivity (4 items), demands at work (12 items), and break (2 items). The sums of the subscales are used, the higher the score, the higher frequency of adverse workstyle practices (i.e., the worse of the outcome).
Self-efficacy | Change from the measurement at baseline (T0) to one week after intervention (T1)
  The exercise self-efficacy will be measured by a 10-item self-efficacy scale with a 4-point-Likert scale (0=completely inaccurate to 3=completely accurate). The higher the score, the higher levels of self-efficacy (i.e., the better outcome)
Mental health | Change from the measurement at baseline (T0) to one week after intervention (T1)
  Mental health will be measured by a 21-item depression, anxiety and stress scale (DASS) with a 4-point Likert scale (0=not applicable and 3 = very often). The higher the score represents a worse outcome.
Body mass index | Change from the measurement at baseline (T0) to one week after intervention (T1)
  Body mass index will be calculated based on the measurement of height (meter) and weight (kilogram) with the formula of kg/m^2. The higher the score represent a worse outcome.
Hip-waist ratio | Change from the measurement at baseline (T0) to one week after intervention (T1)
  Hip-waist ratio will be calculated based on the measurement of hip and waist circumferences (inches) with the formula of waist circumference / hip circumference. The higher the score represents the worse outcome.
Blood pressure | Change from the measurement at baseline (T0) to one week after intervention (T1)
  Blood pressure will be measured by both systolic and diastolic blood pressure. The higher the systolic pressure represents a worse outcome. Also, the higher the diastolic pressure represents a worse outcome.
Social support and exercise | Change from the measurement at baseline (T0) to one week after intervention (T1)
  Social support and exercise will be measured by a 10-item scale with 5-point Likert scale (0=never, and 4=very often). The sum score will be used, the higher the score represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kin Cheung, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Residents Mutual Help Centre, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No